CLINICAL TRIAL: NCT07223970
Title: Target Safety: a Collaboration of Firearm Retailers and Health Care to Address Suicide Prevention
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Sandra L. McKay, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HSC-MS-25-0401
Record Dates: First submitted 2025-10-30; First posted 2025-11-03 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Firearm Injury; Suicide Due to Use of Firearm
Keywords: temporary out-of-home storage (TOHS).

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Temporary out-of-home storage (TOHS) training (Experimental)
  Interventions: Behavioral: Temporary out-of-home storage (TOHS) training

INTERVENTIONS:
Behavioral: Temporary out-of-home storage (TOHS) training — The intervention will consist of a brief conversation with the firearm owner, which will include asking about their planned storage practices, providing education on secure storage options, assessing their knowledge about TOHS, and providing subsequent education about TOHS. The intervention is designed to be brief and conversational, taking no more than 5 minutes. The conversation will be guided by a brochure developed by our expert team, and firearm owners will be directed to additional resources for further information

SUMMARY:
The purpose of the study is to understand how culturally competent messaging on secure firearm storage and temporary out-of-home storage (TOHS) is perceived and accepted by firearm owners.

ELIGIBILITY:
Inclusion Criteria:

* Gun store owners, firearm range owners, and healthcare providers in the greater Houston area

Exclusion Criteria:

* Non-English or Spanish speakers

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability of TOHS education as assessed by the likert scale on the post educational survey | post intervention (about 6 weeks after baseline)
  The survey will be reported categorically as Not at all, Slightly, Moderately, Very, and Extremely

SECONDARY OUTCOMES:
Appropriateness of the intervention's venue (i.e., location for storage services) as assessed by the post educational survey | post intervention (about 6 weeks after baseline)
  There are 3 questions and each is reported categorically as yes or no
Likelihood to talk to family and friends about TOHS as assessed the post educational survey | post intervention (about 6 weeks after baseline)
  This is a 2 item questionnaire and each will be categorically reported as yes or no
Adoptability of TOHS by firearm owners as assessed by the likert scale on the post educational survey | post intervention (about 6 weeks after baseline)
  This will be reported categorically as Strongly Disagree, Disagree, Neutral, Agree or Strongly Agree

CONTACTS AND LOCATIONS:
Overall Officials: Sandra McKay, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No